CLINICAL TRIAL: NCT02893657
Title: The Role and Dynamics of Liver Dysfunction in Patients Undergoing Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Semmelweis University Heart and Vascular Center (Other)
Collaborators: Semmelweis University (Other)
Responsible Party: Principal Investigator, Andrea Szekely, associate professor, Semmelweis University
Other Study IDs: SE AITK VSZÉK LIVER
Record Dates: First submitted 2016-08-30; First posted 2016-09-08 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Cardiac Surgery; Hepatic Impairment; Heart Failure
Keywords: MELD score; hemodynamics; liver abnormalities
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the present study is the evaluation of the occurrence and effect of hepatic dysfunction on outcome following cardiac surgery, as well as the monitoring of changes in liver haemodynamics in the early postoperative period.

DETAILED DESCRIPTION:
Prospective, consecutive study of patients undergoing cardiac surgery in Heart and Vascular Center, Semmelweis University, Budapest.

Registered data:

* Anamnestic and demographic data
* Liver dysfunction prior surgery, etiology of liver dysfunction
* Perioperative clinical data: laboratory tests, imaging, haemodynamic measures
* risk prediction score of the American Society of Anesthesiologists(ASA), EUROpean System for Cardiac Operative Risk Evaluation (EuroScore), Acute Physiology and Chronic Health Evaluation II (APACHE II), Simplified Acute Physiology Score (SAPS II), Canadian Cardiovascular Society grading of angina pectoris (CCS)
* Model for End-Stage Liver Disease (MELD), MELD excluding International Normalised Ratio (INR) (MELD-XI), modified MELD score (modMELD), Child-Pugh

The occurrence and etiology pattern of hepatic impairment are going to be evaluated according to age and type of cardiac illness. Correlations between perioperative haemodynamical alterations and structural, functional changes in hepatic status will be investigated.

The impact of hepatic impairment on surgical outcome is going to be examined by multivariate regression models.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age admitted for elective cardiac surgical procedures

Exclusion Criteria:

* Not willing to participate.
* Pregnant women.
* During active psychiatric hospital care.
* Patients with defined legal incapability or limited capability.
* Non-evaluable patient due to insufficient clinical information
* Patients with a transplanted heart.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cardiac surgical patients
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
The composite of in-hospital death of any cause | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Length of hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Length of ICU stay | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks

SECONDARY OUTCOMES:
Evidence of clinically definite postoperative decline in hepatic function | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Need for reoperation due to bleeding or cardiac cause | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Evidence of clinically definite postoperative pulmonary or systemic congestion | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Evidence of clinically definite postoperative low cardiac output syndrome | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Evidence of clinically definite postoperative acute kidney injury and the need for dialysis | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Evidence of clinically definite postoperative impaired coagulation | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Enikő Holndonner-Kirst, MD, Principal Investigator — Semmelweis University; Andrea Székely, MD, PhD, Study Director — Semmelweis University; Daniel Lex, MD, Principal Investigator — Semmelweis University; Nikoletta Ráhel Czobor, MD, Principal Investigator — Semmelweis University; Ádám Nagy, MD, Principal Investigator — Semmelweis University; János Gál, MD, PhD, Study Chair — Semmelweis University; Béla Merkely, MD, PhD, Study Chair — Semmelweis University
Locations (1):
- Heart and Vascular Center, Semmelweis University, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No